CLINICAL TRIAL: NCT04731545
Title: Evaluation of the Buccal Bone Resorption in Immediate SLActive Implant Placement in Thin vs. Thick Buccal Bone Plates: RCT
Brief Title: Buccal Bone Resorption in Immediate SLActive Implant Placement Thin vs. Thick Buccal Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Hani Elnahass, Assitant Professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 333
Record Dates: First submitted 2021-01-25; First posted 2021-02-01 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Dental Implant; Immediate Implant
Keywords: immediate implant; esthetic zone; buccal plate; SLActive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- thin buccal bone (Active Comparator)
  Interventions: Device: immediate implant placement
- thick buccal bone (Active Comparator)
  Interventions: Device: immediate implant placement

INTERVENTIONS:
Device: immediate implant placement — Minimally traumatic tooth extraction, immediate implant placement and hard tissue grafting. loading after 3 months.

SUMMARY:
The utilization of SLActive implants which allow more rapid osseointgeration with 3 to 4 weeks. will be placed in thin buccal bone as immediate implants to determine the resorption compared to thick buccal bone

DETAILED DESCRIPTION:
With the increased demand for aesthetics and the expectation of immediate tooth replacement, improving the treatment options in case with hopeless teeth in the esthetic zone by immediate implants is a need by both practitioners and patients.

Current guidelines, today, restricting such treatment to only thick (+ or = 1mm) buccal bone plates. However, the literature shows that less than 10% of the community have such criteria, making it a high risk but needed procedure.

Soft tissue and bone remodelling after extraction is an inescapable fact. Immediate implant placement cannot prevent soft tissue and bone remodeling around implants (Araújo et al. 2005, Chen et al. 2009), but implant surface treatment and modifications might enhance the maintainability of the supporting structures around the dental implant due to its faster integration, better stimulating the vascular components at the site. This could be tested by the crestal and buccal bone changes, pink esthetic score and ostell readings.

ELIGIBILITY:
Inclusion Criteria:

1. Single bounded irrestorable tooth in the esthetic zone that needs to be extracted.
2. Healthy systemic condition.
3. Type I socket with a minimum of 1mm of buccal bone thickness prior to extraction. (Morton et al., 2014)
4. Sufficient bone apical to the socket for implant primary stability. (Morton et al., 2014)
5. Good oral hygiene.
6. Patient accepts a minimum of three-year follow-up period (cooperative patients).

Exclusion Criteria:

1. Signs of acute infection related to the area of interest.
2. Patients with parafunctional habits (Lobbezoo et al. 2006 and Roelhing et al. 2016).
3. Smokers (Lambert et al. 2000).
4. Pregnant females.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Bucccal bone changes | 12 months post loading
  standardized Cone beam computed Tomography The radiograph will be taken preoperatively and 12 month after. The pre and post operative cone beams will be compared to each other observing any changes of the buccal bone at 2 , 4 and 6 mm from the crest, the measurements will be in mm

SECONDARY OUTCOMES:
Implant stability | 3 months
  Ostell readings in isq (range from 55 till over 70) bleow 55 low stability over 55 till 65 moderate stability above 70 good stability
Crestal bone changes | 12 months post loading
  Periapical radiograph the measurements will be taken from the platform of the implants. 3 readings will be taken one at the paltform one above and one below according to pattern and form of the resorption.
Soft tissue thickness | 3 months
  Periodontal probe
Post operative pain and swelling | 1 week
  Blinded assessment ( numerical score)
Buccal bone thickness | 3 months
  Cone Beam Computed Topography
Postsurgical satisfaction | 1 week
  Questionnaire
Pink aesthetic score | 12 months post loading
  Pink esthetic score Scale 0 being the lowest and 14 highest attainable

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] ElNahass H, Tawfik OK, Naiem SN, Zazou N, Moussa M. Evaluation of buccal bone resorption in immediate implant placement in thin versus thick buccal bone plates: An 18-month follow-up prospective cohort study. Clin Implant Dent Relat Res. 2024 Jun;26(3):532-544. doi: 10.1111/cid.13312. Epub 2024 Feb 21. PMID 38380779